CLINICAL TRIAL: NCT04333017
Title: Percutaneous Radiofrequency Ablation of Parietal Endometriosis : a Pilot Study (PRFA)
Brief Title: Percutaneous Radiofrequency Ablation of Parietal Endometriosis (PRFA)
Acronym: PRFA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 69HCL19_0826; 2020-A00320-39 (Other: ANSM)
Record Dates: First submitted 2020-03-11; First posted 2020-04-03 (Actual); Last update posted 2025-08-08 (Actual); Status verified 2025-08

CONDITIONS: Endometriosis
Keywords: Parietal endometriosis; Abdominal Wall endometriosis; Percutaneous radiofrequency ablation
MeSH Terms: conditions — Endometriosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- treated patient (Experimental): Percutaneous radiofrequency ablation of parietal endometriosis
  Interventions: Device: Percutaneous radiofrequency ablation of parietal endometriosis

INTERVENTIONS:
Device: Percutaneous radiofrequency ablation of parietal endometriosis — Treatment is carried out under local anaesthesia after surgical asepsis, in interventional radiology room. Radiofrequency needles are inserted percutaneously under ultrasound guidance. Number of needles depends on the size of lesion (1 or 2 or 3 needles). In case of proximity between lesion and peritoneum, artificial ascites can be performed. Treatment is carried out in accordance with device's instructions for use (thyroid nodules treatment algorithm), with a gradual increase in power every 5 minutes, without exceeding the maximum authorised power (depending on number and length of needles). State of coagulation is monitored under visual ultrasound control of ablation area (diffusion of Co bubbles), until a decrease in effective power is obtained. Several ablation zones are performed on the same nodule with overlapping of the different impacts. An ice pack is applied to the treated area. An analgesic PO treatment of step 1 and/or 2 is prescribed for 5 days.

SUMMARY:
Parietal endometriosis is the implantation of endometrial tissue in abdominal structures more superficial than the peritoneum. It is a rare form of the disease (incidence estimated between 0.04 and 12% among women operated on for endometriosis depending on the series) but is classically resistant to medical treatment and can be disabling. Surgical resection is currently the reference treatment in the event of failure of hormonal treatment, despite the sometimes significant skin scars and the risk of parietal fragility that may require a cure of venting by parietal prosthesis. The recurrence rate after surgical resection is 4.3%. The use of radiofrequency for therapeutic purposes is nowadays described in multiple applications such as cardiac arrhythmia, neurological and spinal disorders, as well as for the treatment of liver, kidney, prostate, breast, lung or skin cancers. Its use has already been reported in the field of benign gynecology with, in particular, demonstrated efficacy in the treatment of uterine fibroids by laparoscopic, trans-vaginal or percutaneous means. There are also large published series on radiofrequency for the treatment of adenomyosis, by the transvaginal and laparoscopic route.

In the context of parietal endometriosis, this would be a minimally invasive, percutaneous treatment. Ultrasound guidance allowing good targeting of the lesions and the procedure would most often be carried out on an outpatient basis and under local anaesthesia. And in case of failure or partial effectiveness, the reference treatment would remain accessible for these patients.

There is only one published case of the use of radiofrequency in parietal endometriosis (case reports). Despite results that seem encouraging in terms of a rapid and prolonged therapeutic effect on symptoms, no further cases or series have been published since.

Our study aims to investigate the feasibility of percutaneous radiofrequency treatment for parietal endometriosis, with the secondary objective of evaluating the safety, efficacy and risk factors for failure of the technique.

10 patients will be treated. For follow-up all patients will have an ultrasound and MRI before treatment, then an ultrasound at 1 month, 3 months and 6 months post-treatment and a second MRI at 6 months post-treatment. The investigators will also evaluate pain and quality of life with specific questionnaires at each visit.

ELIGIBILITY:
Inclusion Criteria:

* Patient over 25 years of age;
* Presenting between 1 and 3 lesions of parietal endometriosis, all accessible to radiofrequency treatment, with a major axis less than 10cm;
* Symptomatic (chronic and/or catamenial pain);
* Histological diagnosis of endometriosis;
* In failure of medical treatment;
* Nodule visible on ultrasound;
* Affiliated with or beneficiary of a social security or similar scheme.
* Having signed an informed consent for participation in the study

Exclusion Criteria:

* Presence of a parietal endometriosis lesion with superficial skin involvement (dermis);
* Presence of other symptomatic extra-parietal endometriosis lesions for which surgical treatment is planned;
* Uncontrolled diabetes, i.e. HbA1c >7% despite well-treated and well-controlled treatment;
* Contraindication to the use of radiofrequency: implanted electronic device, such as a pacemaker or self-synchronizing defibrillator; weakened immune system; coagulation disorder;
* Contraindication to the use of Sonovue
* Contraindication to the use of gadolinium
* Severe renal failure (glomerular filtration rate less than 30 ml / min / 1.73m²)
* Pregnant patient or with a desire to become pregnant within 6 months after treatment;
* Patient who is not fluent in the English language;
* Patient over the age of majority protected by law, under curatorship or guardianship;
* Person deprived of liberty by a judicial or administrative decision, person subject to psychiatric care and people admitted to a health or social establishment for purposes other than that of research.
* Patient participating in other interventional research that may interfere with the present research (at the discretion of the investigator);
* Patient who has participated in other research that includes an ongoing opt out period.

Min Age: 25 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2020-06-12 (Actual); Primary Completion 2022-07-27 (Actual); Study Completion 2023-01-31 (Actual)

PRIMARY OUTCOMES:
Feasibility of PRFA. Evaluation by composite criteria with the need to validate all the criteria for the procedure to be considered "feasible". | The day of the treatment (Day 0) - no earlier than 7 days after the 1st visit
  The treatment is considered "feasible" if it meets all of the following criteria:
  * Visualization of the lesion intraoperatively by percutaneous ultrasound (yes/no),
  * Visibility of the posterior aponeurosis/peritoneum interface behind the lesion (yes/no),
  * Placement of one or more radiofrequency (RF) needles within the target lesion (yes/no),
  * Procedure for firing without anomaly (yes/no) :
    * Performing one or more treatment zones until a drop in effective power is obtained, automatically interrupting needle activity and demonstrating the effectiveness of the treatment.
    * complete covering of the nodule by the CO bubbles released by the procedure.

SECONDARY OUTCOMES:
Security and tolerance of PRFA | From the 1st visit (no later than 7 days before treatment (Day -7)) until the end of the study (Month 6)
  Number, type and severity of adverse events related to radiofrequency treatment. Pain during treatment.
radiological effectiveness measured by ultrasonography with Sonovue (composite criteria) | 1 month post therapeutic (Month 1)
  * Diameters (largest, orthogonal to the largest diameter and anteroposterior diameter [in cm]) and volume (in cm3) of the lesions,
  * Echogenicity to muscle (hypo- / iso- / hyper-echoic)
  * Presence of a posterior shadow cone (yes/no)
  * Sonovue characteristics (no, moderate or frank enhancement)
  * US Doppler characteristics (no, slight or marked vascularization)
  * Characteristics in Shearwave elastography (in kPa)
  * Evaluation by the radiologist of the percentage of nodule volume presenting a change in appearance on ultrasound (0% / < 50% / > 50% / 100%)
radiological effectiveness measured by ultrasonography with Sonovue (composite criteria) | 3 month post therapeutic (Month 3)
  * Diameters (largest, orthogonal to the largest diameter and anteroposterior diameter [in cm]) and volume (in cm3) of the lesions,
  * Echogenicity to muscle (hypo- / iso- / hyper-echoic)
  * Presence of a posterior shadow cone (yes/no)
  * Sonovue characteristics (no, moderate or frank enhancement)
  * US Doppler characteristics (no, slight or marked vascularization)
  * Characteristics in Shearwave elastography (in kPa)
  * Evaluation by the radiologist of the percentage of nodule volume presenting a change in appearance on ultrasound (0% / < 50% / > 50% / 100%)
radiological effectiveness measured by ultrasonography with Sonovue (composite criteria) | 6 month post therapeutic (Month 6)
  volume (in cm3) of the lesions,
  * Echogenicity to muscle (hypo- / iso- / hyper-echoic)
  * Presence of a posterior shadow cone (yes/no)
  * Sonovue characteristics (no, moderate or frank enhancement)
  * US Doppler characteristics (no, slight or marked vascularization)
  * Characteristics in Shearwave elastography (in kPa)
  * Evaluation by the radiologist of the percentage of nodule volume presenting a change in appearance on ultrasound (0% / < 50% / > 50% / 100%)
radiological effectiveness measured by MRI with Gadolinium (composite criteria) | 6 month post therapeutic (Month 6)
  * Diameters (largest, orthogonal to the largest diameter and anteroposterior diameter [in cm]) and volume (in cm3) of the lesions
  * signal in T2 sequence with respect to the muscle (hypo- / iso- / hyper-signal) ;
  * presence of T1 hypersignal (yes/no);
  * minimum and maximum ADC (Apparent Diffusion Coefficent) value (in mm²/s);
  * lesional enhancement in the center (yes/no);
  * Peri-lesional enhancement (yes/no);
clinical efficiency (composite criteria) | 1 month post therapeutic (Month 1)
  Assessment of pain related to the lesion: maximum EVA during menstruation and maximum EVA outside of menstruation
clinical efficiency measured by SF36 | 1 month post therapeutic (Month 1)
  Quality of life of patients measured by validated questionnaire in endometriosis: SF36 (Short Form (36) Health Survey)
clinical efficiency measured by EHP-5 | 1 month post therapeutic (Month 1)
  Quality of life of patients measured by validated questionnaire in endometriosis: EHP-5 (Endometriosis Health Profile)
clinical efficiency (composite criteria) | 3 month post therapeutic (Month 3)
  Assessment of pain related to the lesion: maximum EVA during menstruation and maximum EVA (Echelle Visuelle Analogique) outside of menstruation
clinical efficiency measured by SF36 | 3 month post therapeutic (Month 3)
  Quality of life of patients measured by validated questionnaire in endometriosis: SF36
clinical efficiency measured by EHP-5 | 3 month post therapeutic (Month 3)
  Quality of life of patients measured by validated questionnaire in endometriosis: EHP-5
clinical efficiency (composite criteria) | 6 month post therapeutic (Month 6)
  Assessment of pain related to the lesion: maximum EVA during menstruation and maximum EVA outside of menstruation
clinical efficiency measured by SF36 | 6 month post therapeutic (Month 6)
  Quality of life of patients measured by validated questionnaire in endometriosis: SF36
clinical efficiency measured by EHP-5 | 6 month post therapeutic (Month 6)
  Quality of life of patients measured by validated questionnaire in endometriosis: EHP-5
population characteristics (composite criteria) | At the 1st visit: up to 7 days before treatment (Day -7)
  age, gestational age, parity, history of caesarean section, history of gynaecological surgery excluding endometriosis, history of endometriosis surgery, age of diagnosis of endometriosis, age of diagnosis of parietal endometriosis.
Feature of PRFA: power of the shot | The day of the treatment (Day 0) no earlier than 7 days after the 1st visit
  Description of the procedure: power (Watt) of the shot
Feature of PRFA: duration of the shot | The day of the treatment (Day 0) no earlier than 7 days after the 1st visit
  Description of the procedure: duration (min) of the shot.
Feature of PRFA: total duration (min) of the procedure | The day of the treatment (Day 0) - no earlier than 7 days after the 1st visit
  Description of the procedure: total duration (min) of the procedure.

CONTACTS AND LOCATIONS:
Locations (1):
- Hospices Civils de Lyon - Hôpital de la Croix Rousse, Lyon, France

REFERENCES:
- [Result] Haquin A, Delacroix C, Rode A, Taconet D, Maissiat E, Boussel L, Dubernard G, Philip CA. Feasibility of Percutaneous Radiofrequency Ablation for Abdominal Wall Endometriosis: A Prospective Pilot Study. J Minim Invasive Gynecol. 2025 Mar;32(3):288-296. doi: 10.1016/j.jmig.2024.10.022. Epub 2024 Oct 26. PMID 39490892